CLINICAL TRIAL: NCT03279068
Title: Electronic Fetal Monitoring With and Without Pattern Interpretation: A Prospective Cohort Study
Brief Title: Electronic Fetal Monitoring With and Without Pattern Interpretation
Status: Terminated | Type: Observational
Why Stopped: Civil unrest in region/country of study
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Abida Hasan, Maternal Fetal Medicine Fellow, University of Illinois at Chicago
Other Study IDs: 2017-0723
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Cardiotocography
Keywords: electronic fetal monitoring
MeSH Terms: interventions — Educational Status; Paper

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without Pattern Interpretation: All women who are admitted for labor at Ayder Referral Hospital in Mekelle, Ethiopia will be asked to participate and a physician will obtain consent. If an indication arises and they are designated to receive EFM per previously established standard practice at Ayder Hospital, then their patient information will be collected. Patients who require EFM will be asked to provide basic health and demographic information, along with collection of information on labor and delivery course, post-partum outcome, and neonatal outcomes. The investigators estimate enrollment of up to 1800 patients which will result in at least 300 patients who will require EFM.
- With Pattern Interpretation: All women who are admitted for labor at Ayder Referral Hospital in Mekelle, Ethiopia will be asked to participate and a physician will obtain consent. If an indication arises and they are designated to receive EFM per previously established standard practice at Ayder Hospital, then their patient information will be collected.
  Their labor will be managed as in Phase 1 except that EFM will be interpreted and managed as per ACOG/FIGO guidelines using paper on which fetal heart tracings will be recorded. All other aspects of their care will proceed as per standard at Ayder Referral Hospital.
  Patients who require EFM will be asked to provide basic health and demographic information, along with collection of information on labor and delivery course, post-partum outcome, and neonatal outcomes. The investigators estimate enrollment of up to 1800 patients which will result in at least 300 patients who will require EFM.
  Interventions: Other: Teaching and EFM Paper

INTERVENTIONS:
Other: Teaching and EFM Paper — Data will be collected for patients receiving EFM without pattern interpretation as the first phase of the study, as this is the current practice at Ayder Hospital. Then, the second phase will involve a week of teaching sessions regarding interpretation and management of EFM as per ACOG and FIGO guidelines. For the third phase of this study, paper will be provided for the use of EFM with pattern interpretation for all patients receiving EFM.
  Other Names: Teaching and Paper
  Groups: With Pattern Interpretation

SUMMARY:
Cesarean section is one of the most common surgeries performed with the intention of optimizing maternal and fetal/neonatal outcomes. One of the major indications for cesarean delivery is "non-reassuring fetal status" (NRFS). Electronic fetal monitoring is used to evaluate and manage women while they are in labor. A fetal heart rate tracing is recorded on paper or electronically and produces a pattern to allow physicians to visually identify fetuses that are at risk for hypoxia and/or acidemia. This practice allows for prompt intervention via intrauterine resuscitation and expedited delivery if deemed necessary. National and international guidelines published by the International Federation of Gynecology and Obstetrics and American College of Obstetrics and Gynecology describe how fetal heart rate patterns obtained with electronic fetal monitoring should be interpreted and managed. In order to interpret fetal heart rate patterns, the ability to visualize a pattern is necessary. This is made possible either by using paper on which the fetal heart rate is recorded or electronic screens with recording systems. In hospitals where continuous fetal heart rate monitoring is available, but paper resources are depleted and electronic screens are not available, an image of the fetal heart rate pattern cannot be produced nor interpreted. Thus, electronic fetal monitoring is used as an incomplete tool has become standard of care for laboring patients.

Historical Western data revealed that implementation of continuous fetal monitoring with pattern interpretation increased rates of cesarean delivery in comparison to intermittent auscultation. However, it is not clear if the inability to interpret a pattern (because of a lack of paper or electronic recording) results in increased or decreased cesarean rates in comparison to pattern interpretation. It is possible that the implementation of pattern interpretation could decrease cesarean delivery rates allowing increased or earlier opportunity for fetal resuscitation for patients with tracing abnormalities which may avert cesarean delivery. The investigators' aim is to assess cesarean delivery rates using electronic fetal monitoring with versus without pattern interpretation in a hospital in a low-middle income country where resources are lacking.

If a decrease in cesarean delivery rate is observed and/or neonatal outcomes are improved, this study may serve as an impetus to encourage electronic fetal monitoring paper-producing companies to subsidize or donate supplies to hospitals in developing countries. Ensuring that fetal status is in fact non-reassuring by fetal heart rate pattern interpretation prior to proceeding with cesarean delivery may decrease the cesarean delivery rate while not compromising fetal outcomes.

DETAILED DESCRIPTION:
"Intrapartum electronic fetal monitoring (EFM) also known as cardiotocography (CTG) is used for most women who give birth in the United States," as per American College of Obstetrics and Gynecology (ACOG) Practice Bulletin 116 - Management of Intrapartum Fetal Heart Rate Tracings. This document regarding recommendations of intrapartum management functions on the assumption that electronic fetal monitoring is being recorded, either on paper or electronically, to allow for interpretation of the pattern of the fetal heart rate over time. In the US, the widespread availability of electronic medical record systems allows continuous visualization of fetal heart tracings. In hospitals that have not transitioned to electronic recording of fetal heart rate tracings, these tracings are continuously recorded on paper. The guidelines put forth by ACOG in Practice Bulletin 116 define how to interpret patterns of fetal heart rates, and furthermore, how to manage patients based on these interpretations by categorizing features of tracings that are concerning vs. reassuring.

The International Federation of Gynecology and Obstetrics (FIGO), of which ACOG is a member, produced several documents in 2015 to address Consensus Guidelines for Intrapartum Fetal Monitoring. The document addressing CTG for an international audience provides the same guidelines for interpretation of fetal heart tracing patterns as ACOG, and very similar recommendations for management based on slightly different categorization terminology. Both the ACOG Practice Bulletin and the FIGO Consensus Guideline addressing intrapartum fetal monitoring describe fetal heart rate patterns including baseline rate, variability, accelerations, and decelerations. Specifically, they address the various types of decelerations, some of which are benign, and others which are ominous for fetal well-being, as well as the importance of variability in assessing fetal well-being. For example, moderate baseline variability reflects the oxygenation of the central nervous system and reliably predicts the absence of ongoing hypoxic injury and metabolic acidemia at the time it is observed.

An alternative method for intrapartum fetal monitoring is via intermittent auscultation (IA). IA is a technique by which the fetal heart rate is appreciated by a stethoscope, fetoscope, or handheld Doppler to assess the fetal heart rate over established periods of time during different stages of labor, but does not produce a continuous numerical output of the fetal heart rate. As such, certain features of a fetal heart rate pattern cannot be evaluated by IA, including fetal heart rate variability or the different types of decelerations. According to the FIGO Guidelines on Intermittent Auscultation, "Based on expert opinion, IA should be recommended in all labors in settings where there is no access to CTG monitors or to the resources necessary for using them. When the resources for CTG monitoring are available, intermittent auscultation may be used for routine intrapartum monitoring in low-risk cases. However, approximately half of the panel members believe that continuous CTG should be the option during the second stage of labor, although there is no direct scientific evidence to support this." In settings where CTG is available, the conditions required to use IA are stringent and even preclude patients who don't deliver within 1 hour of pushing. Furthermore, management of abnormal findings on IA includes proceeding to CTG if it is available. These provisions to using IA convey the implication that it is preferred to have CTG available for use, if possible. It is important to note that electronic fetal monitoring without paper or the ability to interpret a pattern, is not the same as IA or electronic fetal monitoring as described above. Therefore, there is no set of guidelines to interpret and manage patients monitored with continuous monitoring without pattern interpretation.

In many developing countries, hospitals have the ability to provide intrapartum electronic fetal monitoring. At Ayder Referral Hospital, a teaching hospital for Mekelle University, labor and delivery is equipped with electronic CTG monitors that display fetal heart rate in real time, and potentially have the ability to record on paper. Secondary to limited number of CTG monitors, EFM is reserved for use for patients who are considered "high risk," and IA is used to monitor patients who are "low risk." "High risk" patients are those who have maternal conditions or fetal conditions that prompt higher level of fetal monitoring, such as pre-eclampsia, history of prior cesarean delivery, or concerns regarding fetal well-being. However, at this hospital, as in many other hospitals in sub-Saharan Africa, paper strip supplies were depleted and have not been replenished. Thus, patients are currently monitored intrapartum with a live feedback of fetal heart rate, but with no ability to interpret fetal heart rate pattern. Management of patients in this setting is based on real-time fetal heart rates that are continuously observed, which is an intermediate entity of fetal monitoring for which there are no established recommendations for management. Neither the ACOG Bulletin nor the FIGO Consensus Guidelines address CTG/EFM without pattern interpretation.

In a setting such as Ayder Referral Hospital in Mekelle, making efforts to minimize the cesarean delivery rate while optimizing neonatal outcomes is paramount for many reasons. In Mekelle, personal and socioeconomic implications of a major surgery such as cesarean delivery are considered seriously, and refusal of cesarean delivery is higher in many developing countries in comparison to resource-rich countries. Furthermore, performance of a cesarean delivery in a patient population that has a high aversion to cesarean delivery puts these patients at risk of avoiding a subsequent delivery in a hospital to avoid a repeat cesarean section, which can have dire consequences. Preventing adverse fetal outcome is equally as important as preventing unnecessary cesarean section, as resources available for neonatal resuscitation are limited in comparison to developed countries.

While there is a lack of data regarding the use of EFM without pattern interpretation, the investigators' hypothesis is that the implementation of EFM with pattern interpretation will result in a decrease in cesarean delivery rates without altering neonatal outcomes. This hypothesis arises from anecdotal experience. Providers at Ayder Referral Hospital and the principal investigator's observation of the intrapartum management on Labor and Delivery noted that several of the cesarean deliveries that occurred may have been averted given the opportunity for intrauterine resuscitation.

This prospective cohort study comparing current standard of care at Ayder Referral Hospital (EFM without pattern interpretation for high risk obstetric patients) with EFM as per ACOG and FIGO recommendations (with pattern evaluation) may reveal a change in cesarean delivery rate and/or neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women who have a singleton pregnancy.
* Women admitted for labor to Ayder Referral Hospital in Mekelle, Ethiopia.
* Pregnant women aged 18 years or older.
* Receiving EFM for intrapartum management.
* Patients assigned to receive EFM will be designated by the current protocol regarding "high risk" vs. "low risk" patients at Ayder Referral Hospital as per discretion of the supervising provider in Labor and Delivery.

Exclusion Criteria:

* Women who are carrying multiple gestation.
* Pregnant women under 18 years of age.
* Low risk women who are undergoing IA.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be pregnant.
Study Population: Women of childbearing age presenting for care at Ayder Referral Hospital in Mekelle, Ethiopia. Most patients are from the Tigray, Afar, or Amahara regions in Ethiopia.
Sampling Method: Non-Probability Sample
Enrollment: 637 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Cesarean delivery rate for non-reassuring fetal status | July 2018

SECONDARY OUTCOMES:
Adverse neonatal outcomes | July 2018
  Neonatal demise before mother's discharge, admission to neonatal ICU, duration of neonatal ICU admission, APGAR <7 at 5 minutes
Cesarean delivery rate | July 2018

CONTACTS AND LOCATIONS:
Overall Officials: Abida Hasan, MD, Principal Investigator — University of Illinois, Maternal Fetal Medicine Fellow
Locations (1):
- Ayder Referral Hospital, Mekelle University, Mek'ele, Tigray, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists. Practice bulletin no. 116: Management of intrapartum fetal heart rate tracings. Obstet Gynecol. 2010 Nov;116(5):1232-40. doi: 10.1097/AOG.0b013e3182004fa9. PMID 20966730
- [Background] Ayres-de-Campos D, Spong CY, Chandraharan E; FIGO Intrapartum Fetal Monitoring Expert Consensus Panel. FIGO consensus guidelines on intrapartum fetal monitoring: Cardiotocography. Int J Gynaecol Obstet. 2015 Oct;131(1):13-24. doi: 10.1016/j.ijgo.2015.06.020. No abstract available. PMID 26433401
- [Background] Lewis D, Downe S; FIGO Intrapartum Fetal Monitoring Expert Consensus Panel. FIGO consensus guidelines on intrapartum fetal monitoring: Intermittent auscultation. Int J Gynaecol Obstet. 2015 Oct;131(1):9-12. doi: 10.1016/j.ijgo.2015.06.019. No abstract available. PMID 26433400
- [Background] Malek J. Responding to refusal of recommended cesarean section: Promoting good parenting. Semin Perinatol. 2016 Jun;40(4):216-21. doi: 10.1053/j.semperi.2015.12.009. Epub 2016 Jan 21. PMID 26803168
- [Background] Ohel I, Levy A, Mazor M, Wiznitzer A, Sheiner E. Refusal of treatment in obstetrics - A maternal-fetal conflict. J Matern Fetal Neonatal Med. 2009 Jul;22(7):612-5. doi: 10.1080/14767050802668698. PMID 19479647
- [Background] Ugwu NU, de Kok B. Socio-cultural factors, gender roles and religious ideologies contributing to Caesarian-section refusal in Nigeria. Reprod Health. 2015 Aug 12;12:70. doi: 10.1186/s12978-015-0050-7. PMID 26265149
- [Background] Ajah LO, Ibekwe PC, Onu FA, Onwe OE, Ezeonu TC, Omeje I. Evaluation of Clinical Diagnosis of Fetal Distress and Perinatal Outcome in a Low Resource Nigerian Setting. J Clin Diagn Res. 2016 Apr;10(4):QC08-11. doi: 10.7860/JCDR/2016/17274.7687. Epub 2016 Apr 1. PMID 27190897
- [Background] Ayres-de-Campos D, Arulkumaran S; FIGO Intrapartum Fetal Monitoring Expert Consensus Panel. FIGO consensus guidelines on intrapartum fetal monitoring: Physiology of fetal oxygenation and the main goals of intrapartum fetal monitoring. Int J Gynaecol Obstet. 2015 Oct;131(1):5-8. doi: 10.1016/j.ijgo.2015.06.018. No abstract available. PMID 26433399
- [Background] Boyle A, Reddy UM, Landy HJ, Huang CC, Driggers RW, Laughon SK. Primary cesarean delivery in the United States. Obstet Gynecol. 2013 Jul;122(1):33-40. doi: 10.1097/AOG.0b013e3182952242. PMID 23743454
- [Background] Ayres-de-Campos D, Arulkumaran S; FIGO Intrapartum Fetal Monitoring Expert Consensus Panel. FIGO consensus guidelines on intrapartum fetal monitoring: Introduction. Int J Gynaecol Obstet. 2015 Oct;131(1):3-4. doi: 10.1016/j.ijgo.2015.06.017. No abstract available. PMID 26433398
- [Background] Visser GH, Ayres-de-Campos D; FIGO Intrapartum Fetal Monitoring Expert Consensus Panel. FIGO consensus guidelines on intrapartum fetal monitoring: Adjunctive technologies. Int J Gynaecol Obstet. 2015 Oct;131(1):25-9. doi: 10.1016/j.ijgo.2015.06.021. No abstract available. PMID 26433402